CLINICAL TRIAL: NCT00000822
Title: A Phase I/II Double-Blind Controlled Trial to Determine the Safety and Immunogenicity of HIV-1 MN rgp160 Immuno AG Vaccine Therapy in HIV-Infected Individuals With Greater Than or Equal to 500/mm3 CD4+ T Cells and 200-400/mm3 CD4+ T Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Immuno-US (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 246/946; 11223 (Registry Identifier: DAIDS ES Registry Number); 11499 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Didanosine; Drug Therapy, Combination; HIV Envelope Protein gp160; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Stavudine; HIV Protease Inhibitors; AIDS Vaccines; Ritonavir; Reverse Transcriptase Inhibitors; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ritonavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Ritonavir
Biological: gp160 Vaccine (Immuno-AG)
Drug: Stavudine
Drug: Didanosine

SUMMARY:
To evaluate the safety and immunogenicity of HIV-1 MN rgp160 (Immuno-AG) in HIV-infected patients. To evaluate the immunogenicity of HIV-1 MN rgp160 immunogen by lymphocyte proliferation, specific antibody responses, and DTH reaction. To describe the durability of the immunogen in patients who respond to the first 7 injections when they are boosted every 8 weeks for an additional 6-12 months [AS PER AMENDMENT 11/12/96: stratum 1 patients only]. To describe the ability of the immunogen to induce a response after an additional 6-12 months of injections among patients who did not respond to the first 7 injections [AS PER AMENDMENT 11/12/96: stratum 1 patients only].

HIV-specific cellular immune responses appear to play an important role in HIV disease progression since both T helper and cytotoxic function against HIV decrease with disease progression.

DETAILED DESCRIPTION:
HIV-specific cellular immune responses appear to play an important role in HIV disease progression since both T helper and cytotoxic function against HIV decrease with disease progression.

Patients with CD4 counts greater than or equal to 500 cells/mm3 are randomized to receive HIV-1 MN rgp160 (Immuno-AG) or control. Patients with CD4 counts 50-499 cells/mm3 receive didanosine (ddI) and are then randomized to receive ddI plus vaccine or control. Vaccine or control is given every 4 weeks for 7 injections, then every 8 weeks for 6-12 months or until 1 year after the last patient is randomized. AS PER AMENDMENT 11/12/96: Stratum 1 is composed of 16 subjects with CD4+ T cells greater than or equal to 500 mm3. These subjects are randomized to vaccine therapy or vaccine control. HIV-1 MN rgp160 vaccine or control is given every 4 weeks for 7 injections (Schedule 1), then every 8 weeks until 52 weeks after the last subject has been randomized to stratum 1 (Schedule 2). Stratum 1 patients receive ddI or d4T only if their CD4 cell count has a sustained decrease on 2 consecutive occasions 10-14 days apart and/or HIV/RNA plasma viral load increases to greater than 10,000 copies/ml on 2 consecutive occasions 10-14 days apart. Stratum 2 is composed of 30 subjects with CD4+ T cells 200-400/mm3; accrual to this stratum was activated based on preliminary results from stratum 1 (closed as of 4/5/97). Patients on stratum 2 (open as of 3/4/97) initially receive ritonavir at escalating doses for 2 weeks. Subjects then have ddI and d4T added to the regimen for 7 weeks. Subjects are then randomized to vaccine therapy or vaccine control every 4 weeks for 7 injections, with ritonavir/ddI/d4T continued during vaccine therapy.

AS PER AMENDMENT 3/23/98: As of 6/1/98 vaccine consists of sodium chloride for injection (USP).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* ddI [AS PER AMENDMENT 11/12/96: and d4T]. (Note:
* Patients in the stratum receiving only vaccine or control may take ddI [AS PER AMENDMENT 11/12/96:
* and d4T] ONLY IF their CD4 counts have shown a sustained decrease on two consecutive occasions 10-14 days apart.)
* PCP prophylaxis.
* Treatment for acute conditions, as indicated.

AS PER AMENDMENT 11/12/96:

* Co-enrollment on other research trials.

Patients must have:

* HIV positivity.
* Asymptomatic disease.
* CD4 count >= 50 cells/mm3 (CD4 count must be 50-499 cells/mm3 in patients receiving ddI plus vaccine or control, and must be >= 500 cells/mm3 in patients receiving vaccine or control only)

[AS PER AMENDMENT 11/12/96:

* CD4 count >= 500 cells/mm3 for stratum 1 patients and 200-400 for stratum 2 patients].
* HLA A2 positive documentation.
* An Epstein Barr virus B cell line established within 90 days prior to study entry.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Study is NOT approved for prisoner participation.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Medical contraindication to study participation or inability to comply with study requirements.
* Grade 2 or worse peripheral neuropathy (applicable only to patients receiving ddI plus vaccine or control).

Concurrent Medication:

Excluded:

* Immunomodulating agents, such as inosiplex, ditiocarb sodium, lithium, interferons, interleukin-2, and systemic steroids.
* Any antiretroviral therapy that may increase the risk of peripheral neuropathy (e.g., stavudine, zalcitabine [AS PER AMENDMENT 11/12/96:
* e.g., zalcitabine or lamivudine]).
* Agents such as IV pentamidine that may increase the risk of pancreatitis.
* Standard of care vaccines (in patients receiving vaccine) [AS PER AMENDMENT 11/12/96:
* Standard of care immunizations are permitted 60 days before Schedule 1 vaccine therapy and during Schedule 2 vaccine therapy (but not within 2 weeks of study immunization)].

AS PER AMENDMENT 11/12/96:

* Rifabutin, disulfiram (antabuse), or other medication with similar effects, including metronidazole.

  6.AS PER AMENDMENT 11/12/96:
* The following are prohibited in patients receiving ritonavir:
* amiodarone, astemizole, bepridil, bupropion, cisapride, clozapine, encainide, flecainide, meperidine, piroxicam, propafenone, propoxyphene, quinidine, rifabutin, terfenadine, alprazolam, clorazepate, diazepam, estazolam, flurazepam, midazolam, triazolam, and zolpidem.

Patients with the following prior conditions are excluded:

* History of grade 2 or worse liver abnormality.
* Known allergy to vaccine components.
* Chronic diarrhea persisting for 4 or more weeks within 30 days prior to study entry.
* History of pancreatitis (applicable only to patients receiving ddI plus vaccine or control). [AS PER AMENDMENT 11/12/96:
* History of chronic pancreatitis or history of acute pancreatitis within 2 years prior to entry (stratum 2 patients only).]

Prior Medication:

Excluded:

* Any prior anti-HIV vaccines.

Excluded within 90 days prior to study entry:

* Immunomodulating agents, such as Inosiplex, ditiocarb sodium, lithium, interferons, interleukin-2, and systemic steroids.
* Any antiretroviral therapy that may increase the risk of peripheral neuropathy (e.g., stavudine, zalcitabine [AS PER AMENDMENT 11/12/96:
* e.g., zalcitabine or lamivudine]).
* Agents such as IV pentamidine that may increase the risk of pancreatitis.
* Any treatment for an AIDS-defining illness (applicable ONLY to patients in the stratum receiving ddI plus vaccine or control).

Excluded within 6 months prior to study entry:

* Any other antiretrovirals or immunomodulators besides those mentioned above.
* Allergy desensitization or other vaccines [AS

PER AMENDMENT 11/12/96:

* excluded within 60 days prior to entry].

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46
Dates: Study Completion 1999-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kundu Smriti, Study Chair; Merigan T, Study Chair
Locations (1):
- Stanford CRS, Stanford, California, United States

REFERENCES:
- [Background] Katzenstein D, Valentine F, Kundu S, Haslett P, Smith G, Merigan T. Delayed-type-hypersensitivity reactions to intradermal gp160 in HIV infected individuals immunized with gp160. Int Conf AIDS. 1992 Jul 19-24;8(2):A35 (abstract no PoA 2192)
- [Background] Kundu-Raychaudhuri S, Sevin A, Kilgo P, Nokta M, Pollard RB, Merigan TC. Effect of therapeutic immunization with HIV type 1 recombinant glycoprotein 160 ImmunoAG vaccine in HIV-infected individuals with CD4+ T cell counts of >or=500 and 200-400/mm3 (AIDS Clinical Trials Group Study 246/946). AIDS Res Hum Retroviruses. 2001 Oct 10;17(15):1371-8. doi: 10.1089/088922201753197033. PMID 11679149